CLINICAL TRIAL: NCT04153175
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Assess Intracerebroventricular (ICV) Delivery of CT-010 Via an Implantable Pump and a Cranial Port and Double Lumen Catheter (ICVRX) in Subjects With Focal Seizures, With Temporal Lobe Onset With or Without Secondary Generalization
Brief Title: Study to Assess Intracerebroventricular (ICV) Delivery of CT-010 in Subjects With Focal Seizures, With Temporal Lobe Onset With or Without Secondary Generalization
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Cerebral Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN100P.01
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CT-010 Active Therapy (Active Comparator): Subjects in the active comparator arm will have been randomized to receive active therapy through the implanted drug delivery system through the 3-month blinded period.
  Interventions: Combination Product: ICV delivery of CT-010 via an implantable pump and a cranial port and dual lumen catheter (CIC)
- Placebo (Placebo Comparator): Subjects in the placebo comparator arm will have been randomized to receive placebo therapy through the implanted drug delivery system for the 3-month blinded period.
  Interventions: Combination Product: Placebo delivery via an implantable pump and a cranial port and dual lumen catheter (CIC)

INTERVENTIONS:
Combination Product: ICV delivery of CT-010 via an implantable pump and a cranial port and dual lumen catheter (CIC) — Subjects will be implanted with a drug delivery pump and catheters leading to the ICV space allowing delivery of CT-010.
  Arms: CT-010 Active Therapy
Combination Product: Placebo delivery via an implantable pump and a cranial port and dual lumen catheter (CIC) — Subjects will be implanted with a drug delivery pump and catheters leading to the ICV space allowing delivery of a placebo (saline).
  Arms: Placebo

SUMMARY:
This is a Phase 2 double-blind, randomized, placebo-controlled study to assess the safety and efficacy of ICV delivery of CT-010 via an implantable pump and a cranial port and dual lumen catheter (CIC) in subjects with focal seizures, with temporal lobe onset with or without secondary generalization. Up to 70 subjects will be enrolled. Eligible subjects will be randomized in a 1:1 ratio to either CT-010 or placebo treatment. Up to 20 clinical centers will be enrolled.

DETAILED DESCRIPTION:
Epilepsy patients that are refractory to oral anti-epileptic drug (AED) treatment have significantly higher mortality, higher morbidity, higher economic costs and diminished quality of life compared to those who suffer from epilepsy that can be adequately controlled with medical management. Current options for refractory patients include neurosurgical brain resection, responsive neurostimulation, and vagal nerve stimulation. None of these options is satisfactory due to the low applicability of surgery for patients with poorly localized or multifocal seizures and the limited success of currently available alternative treatment options.

In this study, patients with medically refractory focal epilepsy will be treated with intracerebroventricular (ICV) administration of CT-010, a reformulation of valproate, using an implantable drug pump system. This is a randomized, double-blind Phase 2 study evaluating the efficacy and safety of this therapy. Clinical assessments, adverse events (AEs), seizure diaries, concomitant medications, blood samples and cerebrospinal fluid (CSF) will be collected and reviewed at designated time points. Magnetic resonance imaging (MRI) and electroencephalography (EEG) will also be performed. Subjects will have their surgery, dose changes and pharmacokinetics performed in an inpatient setting.

Subjects will be enrolled based on Inclusion/Exclusion Criteria and undergo a 6-week baseline period confirming and establishing monthly seizure rate. Following the baseline period subjects will undergo system implant and a 1-month implant recovery period. Following successful implant and recovery subjects will be randomized to either active therapy or placebo for a 3-month blinded evaluation period. At the conclusion of the blinded evaluation period, subjects will roll into an Open Label Extension Period, CLN100P.02. Subjects that were randomized to placebo will receive active therapy during CLN100P.02.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

-

For a subject to be eligible for this study, he or she must meet ALL of the following criteria:

1. Subject is male or female between the ages of 18 to 70 years old.
2. Subject is considered an appropriate surgical candidate by the implanting Neurosurgeon.
3. Subject has had confirmed refractory epilepsy for a minimum of 2 years, with unilateral or bilateral temporal lobe involvement with no more than 2 known extratemporal foci.
4. In the opinion of the Investigator, subject has disabling seizures.
5. Subject has had at least one seizure recorded by EEG or video EEG or invasive monitoring within the past 3 years consistent with focal temporal lobe seizures (a normal interictal EEG is consistent with focal seizures)
6. Subject has not achieved effective results previously from at least 3 AEDs in single or combination. An AED may be counted as failed medication if subject has been on it for at least 3-months and is still refractory.
7. Subject failed to obtain an adequate intake of oral valproate of at least 1,000 mgs a day and/or to achieve serum level of at least 60 µg/mL or in the opinion of the Investigator is not a candidate for oral valproate (including subject preference)
8. Per medical history, for the 3 months before informed consent an average of six or more disabling focal seizures of temporal lobe onset, with or without secondary generalization, per month.
9. Subject has seizures that are distinct, stereotypical events that can be reliably counted, in the opinion of the Investigator, by the subject or caregiver.
10. Subject understands study procedures and has voluntarily provided signed, informed consent in accordance with institutional and local regulatory requirements.
11. Subject agrees to maintain the diary for the duration of the study alone or with the assistance of a competent individual.

Subjects must NOT meet any of the following Exclusion criteria to be eligible for enrollment:

1. Subject has any neurologic or medical disease that is likely to progress over the course of the study and/or would interfere with the study.
2. Subject has any coagulopathy, ventricular anatomic distortion, or previous brain resection.
3. Subject has history, within 12 months prior to consent, of repetitive seizures that cannot be counted with confidence by the subject or competent adult/caregiver.
4. Subject has history of psychogenic nonepileptic seizures or seizures secondary to illicit drug or alcohol use, neoplasia, active central nervous system infection, demyelinating disease, degenerative neurological disease, progressive CNS disease or metabolic illness.
5. Subject has had status epilepticus refractory to benzodiazepines and a second agent within one year prior to consent
6. Subject is currently taking neuroleptic medication for behavior control.
7. Subject has a clear brain anatomic structural related lesion which distorts the normal anatomy or interferes with CSF fluid flow.
8. Subject has required (in addition to low dose stable use of benzodiazepines as part of antiepileptic regimen), in the 3 months prior to consent, benzodiazepine use more than 5 times per month for rescue seizure control. One use is defined as taking up to 3 doses in a 24-hour period.
9. Subject is currently implanted with an activated DBS, or RNS device used for treatment of a neurologic or psychiatric condition.
10. Subject currently has VNS and the VNS stimulation parameters are not stable. Stable shall be defined such that the stimulation parameters have not been changed in the last 3 months or the patient/designee is able to report "magnet swipe" during the same time period. The Investigator believes that the continued stable parameters can be maintained through the Primary Evaluation Period.
11. Subject has had more than 10 seizures in one day or more than 200 seizures in one month within last year.
12. Subject has known allergy to citrate, citric acid, valproic acid, divalproex sodium, any components of CT-010, or Depacon®.
13. Subject has unstable depression being treated with more than 1 antidepressant medication or has current evidence of or history within the past 2 years of DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, and has had a suicide attempt within the previous five years. Also excluded are subjects with a history of prolonged postictal psychosis or psychosis or depression secondary to a discontinued AED.
14. In the opinion of the Investigator, the subject has a clinically significant or unstable medical condition (e.g., uncontrolled diabetes or CHF) or a progressive CNS disease that would limit the subject's entry into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Median frequency of total monthly seizures during the Primary Evaluation Period as compared to the Baseline Period as well as a comparison of this Baseline Period/Primary Evaluation Period ratio for the active vs. placebo treatment groups | 84 days

SECONDARY OUTCOMES:
Seizure Severity Questionnaire (SSQ) | 84 days
  Evaluation of change in seizure severity during the blinded period by evaluating any change in the SSQ scores between baseline and Day 84 of blinded period where a lower score is an improvement in condition.
QOLIE-10 | 84 days
  Evaluation of change in quality of life during the blinded period by evaluating change in QOLIE-10 scores between baseline and 84-day evaluations.
Patient Global Impression of Change (PGIC) | 84 days
  Evaluation of subjects impression of therapy efficacy through the PGIC questionnaire at the conclusion of the blinded period. Scale is a single question with a score of 1-7 with a higher score representing a greater improvement in condition. The score is also captured as a VAS of 1-10 again with a higher score representing a greater improvement in condition.
BDI | 84 days
  Evaluation of depression through the BDI questionnaire
BAI | 84 days
  Evaluation of anxiety through the BAI questionnaire

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (7):
  - Mater Hospital Brisbane, Brisbane, New South Wales
  - RBWH, Brisbane, New South Wales
  - Royal Brisbane Medical Center, Brisbane, New South Wales
  - The Mater, Brisbane, New South Wales
  - SVHM, Melbourne, Victoria
  - The Alfred, Melbourne, Victoria
  - The Austin, Melbourne, Victoria
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No